CLINICAL TRIAL: NCT07247890
Title: Research on the Development and Application of a Preoperative Assessment Model for Transcatheter Mitral Valve Edge-to-Edge Repair Based on Visual Foundation Models
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025BJYYEC-KY205-01
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Mitral Regurgitation (MR)
Keywords: Mitral regurgitation (MR); Transcatheter Mitral Valve Edge-to-Edge Repair; Vision Mamba; Visual Foundation Model
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Model Construction, Validation, and Optimization — Data from patients in this study will be used for model construction, validation, and optimization.

SUMMARY:
Mitral regurgitation (MR) is the most prevalent valvular heart disease in China. Transcatheter edge-to-edge repair (TEER) is currently the preferred treatment for patients with severe MR who face high surgical risks. However, existing preoperative assessment methods for TEER suffer from numerous limitations, including complex measurement parameters, high technical demands, and significant subjectivity. Vision Mamba, a cutting-edge technology in the visual domain, overcomes the limitations of common computational units in convolutional neural networks and Transformers through bidirectional state space models and positional encoding, demonstrating exceptional performance in visual tasks. To date, no studies have applied Vision Mamba to ultrasound videos for constructing TEER preoperative assessment models. Our team previously established a Transformer-based evaluation model using a small, single-center cohort. This study innovatively introduces a Vision Mamba-based visual foundation model. By integrating multi-faceted, multi-modal ultrasound videos from multiple centers, we develop a one-stop preoperative TEER assessment model for MR patients [slice identification → video analysis → multi-modal information fusion → preoperative assessment recommendation (suitable/challenging/unsuitable)]. This model will optimize surgical patient identification and accurately screen patients with contraindications. Furthermore, the one-stop model is fast and objective, significantly improving clinical efficiency. It holds promise for deployment at primary care levels to optimize healthcare resource allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-90 years
2. Patients with moderate to severe or severe mitral regurgitation as indicated by echocardiography

Exclusion Criteria:

1. Moderate or severe aortic stenosis or aortic regurgitation, or following aortic valve replacement
2. Patients with congenital heart disease
3. Poor image quality: Insufficient cross-sectional coverage or inability to perform effective mitral valve marking

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was drawn from Beijing Hospital and Fuwai Hospital of the Chinese Academy of Medical Sciences.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Echocardiography-related indicators | Echocardiogram within 2-3 days after admission

IPD SHARING:
Plan to Share IPD: No